CLINICAL TRIAL: NCT01321268
Title: Safety and Efficacy of an Antioxidant Based Dietary Supplement With PUFAs in Healthy Female Volunteers With Cellulite (Orange Peel Skin)
Brief Title: Safety and Efficacy of a Dietary Supplement in Females With Cellulite
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: sponsor stopped study due to recruitment problems
Sponsor: DSM Nutritional Products, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2009-11-03-CEL
Record Dates: First submitted 2011-03-10; First posted 2011-03-23 (Estimated); Last update posted 2015-06-08 (Estimated); Status verified 2012-02

CONDITIONS: Cellulite (Orange Peel Skin)
Keywords: orange peel skin; cellulite
MeSH Terms: conditions — Cellulite | interventions — Dietary Supplements; Fatty Acids, Unsaturated; Resveratrol; Lycopene; beta Carotene; Lutein

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- dietary supplement for cellulite (Experimental): PUFA, resveratrol, lycopene, beta carotene, lutein
  Interventions: Dietary Supplement: dietary supplement for cellulite (PUFA, resveratrol, lycopene, beta carotene, lutein)
- Control (Active Comparator): Vitamin E
  Interventions: Dietary Supplement: Viatmin E

INTERVENTIONS:
Dietary Supplement: dietary supplement for cellulite (PUFA, resveratrol, lycopene, beta carotene, lutein) — oral, twice daily in morning and evening for 6 months
  Arms: dietary supplement for cellulite
Dietary Supplement: Viatmin E — oral, twice daily in morning and evening for 6 months
  Arms: Control

SUMMARY:
To investigate the safety and efficacy of a dietary supplement on cellulite alleviation, fat deposits and quality of life.

DETAILED DESCRIPTION:
The study will be conducted as a single centre, randomized, double-blind, controlled, parallel group study with healthy female volunteers, aged 18-45 years of age, with skin phototypes I to VI and a clinical diagnosis of cellulite on buttocks (at least score 6 at Cellulite Severity Scale (CSS)).

The study will take 24 weeks (6 months) per subject. There will be one previsit during the screening phase and 8 visits per subject during the treatment phase.

Safety and efficacy variables will be performed monthly.

ELIGIBILITY:
Inclusion Criteria:

* Healthy female volunteers
* Age between 18 and 45 years at Day 01 of the study
* Body mass index (BMI) from 18.5 -24.9
* All Fitzpatrick skin types
* CSS score of at least 6
* Normal eating habits (no vegetarians or vegans)
* Written informed consent

Exclusion Criteria:

* Menopause and pre-menopause
* Smoking
* Pregnant women or women intending to become pregnant during study
* Lactation period
* Any kind of dermatological conditions
* Vegetarians or vegans
* Any kind of hepatitis, including any alteration in transaminases
* Use of illicit drugs
* Other surgical or internal diseases e.g. a metabolic or endocrine disease that may affect the outcome of the study (e.g. diabetes, liver diseases, kidney disorders) or having a history of medical or surgical events that may significantly affect the study outcome including any cardiovascular disease, skin disease, hypertension (>160/95 mm Hg at repeated measurements)
* Existence of scars and/or pigmentation in measurement areas (thighs and buttocks), which can influence study measurements
* Participation in any other clinical trial including blood sampling and/or administration or substances up to 30 days before Day 01 of this study
* Any prior aesthetic surgery (Liposuction, Subcision®), 3 months before the study, that may interfere with results
* Any other prior anti-cellulite treatment or body measures treatment, 30 days prior to the study
* Participation in any other non-invasive clinical trial up to 30 days before Day 01 of this study, including blood sampling
* Recent blood or plasmapherese donation (less than 1 month prior to Day 01 of the study)
* Under medical treatment for a skin disease in the past and/or present with a therapy, which may influence the results of the study (systemic steroids or antibiotics, local steroids or topical immunomodulators during the last 3 months
* Use of sun beds or self-tanning products or sun exposure for one month before and during study
* Not willing to accept information-transfer concerning participation in the study, or information regarding his/her health, like laboratory results, findings at anamnesis or physical examination and eventual adverse events to and from his general practitioner
* Subjects intending to initiate any intensive sports
* Every other condition that the investigator might consider to involve a risk for the study subject.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2011-05; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Clinical biochemistry (hematology, blood chemistry, blood coagulation) | 6 months
  change in clinical biochemistry at 6 months vs baseline
vital signs | 6 months
  change in clinical examination at 6 months vs baseline
adverse events and tolerability | 6 months
  change in number of persons with adverse events at 6 months vs baseline

SECONDARY OUTCOMES:
cellulite severity | Day 1, 7, 30, 60, 90, 120, 150, 180
  change in cellulite severity grading according to the cellulite severity scale (CSS)(visual morphological aspects) within repeated measurements
Thigh circumference | Day 1, 7, 30, 60, 90, 120, 150, 180
  Change in thigh circumferences below gluteus fold within repeated measurements, Change in thigh circumferences above the upper part of the knee within repeated measurements
Digital photography | Day 1, Day 90, Day 180
  Change in digital photography Day 90 vs Day 1 Change in digital photography Dag 180 vs Day 1
Ultrasound sonography | Day 1, Day 90 and Day 180
  Change in ultrasound Day 180 vs Day 1, Change in ultrasound Day 90 vs Day 1
Magnetic resonance | Day 1 and Day 180
  change in adipose tissue Day 180 vs Day 1
satisfaction questionnaire | Day 1, Day 30, Day 60, Day 90, Day 120, Day 150, Day 180
  Improvement in patient satisfaction
dermatology life quality index | day 1, 30, 60, 90, 120, 150, 180
  Improvements in the parameters of quality of life
celluquol questionnaire | day 1, 30, 60, 90, 120, 150, 180
  each question in repeated measurements
cutometry | day 1, 90, 180
  change in skin elasticity from day 180 to day 1, change in skin elasticity from day 90 to day 1
corneometry | day 1, 90, 180
  change in skin hydration day 180 vs day 1, change in skin hydration day 90 vs day 1
skin profilometry | day 1, 90, 180
  change in skin topography day 180 vs day 1, change in skin topography day 90 vs day 1
liquichip analysis | day 1, day 180
  change in inflammatory markers day 180 vs day 1

CONTACTS AND LOCATIONS:
Overall Officials: Doris M Hexsel, MD, Principal Investigator — Brazilian Center for Studies in Dermatology (CBED)
Locations (1):
- CBED: Brazilian Center for Studies in dermatology, Porto Alegre, Rio Grande do Sul, Brazil